CLINICAL TRIAL: NCT01184209
Title: Prospective Cohort-study on the Incidence of Adrenal Crisis in Patients With Chronic Adrenal Insufficiency
Brief Title: Prospective Study on the Incidence of Adrenal Crisis in Patients With Chronic Adrenal Insufficiency
Status: Completed | Type: Observational
Sponsor: University of Wuerzburg (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Bruno Allolio, MD, University of Wuerzburg
Other Study IDs: WueAC17/07
Record Dates: First submitted 2010-08-17; First posted 2010-08-18 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2014-01

CONDITIONS: Adrenal Insufficiency
MeSH Terms: conditions — Adrenal Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Prospective study to evaluate incidence, causes and potential risk factors for adrenal crisis in patients with chronic adrenal insufficiency.

DETAILED DESCRIPTION:
This is a prospective study following patients with chronic adrenal insufficiency by contacting them every 6 months via questionnaires and telephone. QUestionnaires assess incidence and causes of adrenal crisis, frequency of hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* chronic primary or secondary adrenal insufficiency requiring glucocorticoid substitution therapy

Exclusion Criteria:

* adrenocortical carcinoma
* long term glucocorticoid treatment above 7.5 mg prednisone equivalent dose for other reasons than adrenal insufficiency
* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients with chronic secondary or primary adrenal failure
Sampling Method: Probability Sample
Enrollment: 444 (Actual)
Dates: Start 2007-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
incidence of adrenal crisis | during study period

SECONDARY OUTCOMES:
mortality | during study period

OTHER OUTCOMES:
hospital admission | during study period

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Allolio, MD, Study Chair — University of Wuerzburg
Locations (2):
- Germany (2):
  - University of Berlin, Berlin
  - University of Wuerzburg, Würzburg

REFERENCES:
- [Derived] Hahner S, Spinnler C, Fassnacht M, Burger-Stritt S, Lang K, Milovanovic D, Beuschlein F, Willenberg HS, Quinkler M, Allolio B. High incidence of adrenal crisis in educated patients with chronic adrenal insufficiency: a prospective study. J Clin Endocrinol Metab. 2015 Feb;100(2):407-16. doi: 10.1210/jc.2014-3191. Epub 2014 Nov 24. PMID 25419882